The Effects of Experiential HIV Testing to Improve
HIV related Knowledge, and Reduce Stigma Toward
HIV of Emergency Department Nurses

| Title | The Effects of Experiential HIV Testing to Improve HIV |
|---|---|
| | related Knowledge, and Reduce Stigma Toward HIV of |
| | Emergency Department Nurses |
| Methodology | Randomized controlled trial |
| Duration of Study | estimated duration for main protocol (from starting of |
| | screening to the last subject processed and finishing the |
| | study) is approximately 4 months. |
| Location of Study | single-center (National Taiwan University Hospital, |
| | Taipei, Taiwan) |
| Objective | improving their knowledge about HIV screening and |
| | reducing their attitudes towards HIV stigma |
| Number of Subjects | 74 completed data. |
| Main inclusion<br>criteria | 1. Age≥20 |
| | 2. clinical nurse working in emergency department |
| | 3. never received an HIV screening due to non- |
| | occupational HIV exposure risk. |
| | 4. no working experience associated with HIV/AIDS, |
| | for example, be a nurse working in an infection |
| | department or as a HIV case manager. |
| | The score as measured by |
| measurement<br>materials | (1) HIV screening knowledge scale(self- |
| | administered) :28 items |
| | (2) Health Care Provider HIV/AIDS Stigma Scale |
| | (translated to Mandarin): 30 items |
| Statistical | the effects of the intervention between the two group |
| | were analyzed by Analysis of Covariance (ANCOVA). |
| Methodology | |
| L | ı |

**Background:** In emergency department (ED) of hospital, human immunodeficiency virus (HIV) testing and/or confirming the patient's HIV status to provide corresponding instructions and answering caregiver's inquiries are conducted frequently due to triage and disease diagnosis process. However, insufficient clinical education and training on HIV-related issues, as well as limited care experience to HIV patients, may lead to fear and HIV-related stigma attitudes among nurses of ED.

**Objectives:** The purpose of this research was to develop an intervention measure of "experiential HIV testing". During the protocol, the nurses of ED directly participated in the complete process of HIV anonymous screening as the role of people who need to be screened, and the consultation contents of HIV testing were provided to them, to verify the following effects: (1) Improving their knowledge about HIV screening (2) Reducing their attitudes towards HIV stigma.

Methods: This study was an experimental research design between November 2022 and February 2023 in an ED of a medical center in Northern Taiwan. The participants were randomly assigned into experimental group and control group. The recruitment criteria included: those who were nurses in ED currently and were performing nursing practices, had no care experiences for AIDS/HIV patients, and had not received an HIV screening due to "non-occupational exposure risk". After signing the written consent form, the pre-test written questionnaires, demographic data sheet, HIV screening knowledge scale, and Health Care Provider HIV/AIDS Stigma Scale (HPASS), were provided to the participants and the data were collected. The experimental group received the intervention of "experiential HIV testing ", which was to give HIV testing kit for self-testing and guide the screening operation process, and to use text teaching materials to deliver HIV pre-test information and post-test consultation services. The subjective opinions of the intervention were also collected of the experimental group. The time of ntervention was about 25-30 minutes; while the control group only accepted the text teaching materials. All post-test were conducted after four weeks for both groups. The data obtained in the study were presented using descriptive statistics, and the effects of the intervention between the two group were analyzed by Analysis of Covariance (ANCOVA).

**Outcome:** It is expected that the intervention "experiential HIV testing" could effectively improve the HIV screening knowledge of nurses of ED, and reduce the stigma attitude towards HIV/AIDS through the role transformation and immersive reflection.

## Flow Chart of the Study

